CLINICAL TRIAL: NCT02965183
Title: The Correlation Between Adenoid Hypertrophy and Body Temperature in Children Before and After Adenoidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Principal Investigator, Itzhak Braverman, Head Otolaryngology Head and Neck Surgery Department, Hillel Yaffe Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0050-15
Record Dates: First submitted 2016-11-13; First posted 2016-11-16 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Otolaryngological Diseases
MeSH Terms: conditions — Otorhinolaryngologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temperature measurements (Experimental)
  Interventions: Other: Temperature measurements

INTERVENTIONS:
Other: Temperature measurements

SUMMARY:
Examination of the correlation between adenoid hypertrophy and body temperature in candidate children for adenoidectomy after exercise

DETAILED DESCRIPTION:
Examination of the correlation between adenoid hypertrophy and body temperature in candidate children for adenoidectomy after exercise.

Adenoid hypertrophy and adenoiditis are accompanied by chronic rhinitis with or without otitis media. It is very common phenomena at ages 2-6 years and those children are symptomatic with snoring, rhinitis, nasal obstruction.

In healthy children with nasal obstruction, body temperature can be elevated following exercise.

As adenoiditis and chronic rhinitis are accompanied by inflammatory process, we would like to examine body temperature of children with adenoid hypertrophy before after exercise.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children with adenoid hypertrophy with or without OSA, SOM Parental concent. No other diseases

Exclusion Criteria:

* Syndromatic children Other diseases If getting antibiotics or other medications

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Changes in temperature | one week before the surgery and one week after the surgery